CLINICAL TRIAL: NCT04328870
Title: The Impact of Spinal Anesthesia and Use of Oxytocin on Fluid Absorption in Patients Undergoing Operative Hysteroscopy; Results From a Prospective Controlled Study
Brief Title: Fluid Absorption in Patients Undergoing Operative Hysteroscopy; Results From a Prospective Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor and Consultant, University of Jordan
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IORG0007981
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Fluid Overload
MeSH Terms: conditions — Edema | interventions — Oxytocin; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin and spinal anesthesia (Active Comparator): spinal anesthesia combined with intravenous oxytocin infusion
  Interventions: Other: oxytocin and spinal anesthesia
- general anesthsia (Active Comparator): general anesthesia alone
  Interventions: Other: General anesthsia

INTERVENTIONS:
Other: oxytocin and spinal anesthesia — start oxytocin 10 IU/200 ml saline at the insertion of the spinal anesthesia
  Arms: oxytocin and spinal anesthesia
Other: General anesthsia — General anesthesia alone.
  Arms: general anesthsia

SUMMARY:
To determine if combining intravenous oxytocin infusion and spinal anesthesia will reduce the amount of glycine absorption in patients undergoing operative hysteroscopy

DETAILED DESCRIPTION:
Prospective controlled study in premenopausal patients who had hysteroscopic surgery including endometrial resection, endometrial polypectomy, myomectomy resection and uterine septal resection. The effect of combined spinal anesthetic with oxytocin infusion on fluid deficit was studied.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal with no cardiovascular comorbidities

Exclusion Criteria:

* endometrial cancer cases, patients who received pre-operative hormonal preparations, previously resected cases and cases done using bipolar diathermy.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pre-menopausal
Enrollment: 88 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
fluid overload | 16 months
  Fluid (glycine) excessive absorption into the patient

CONTACTS AND LOCATIONS:
Overall Officials: Abdelkarim ALoweidi, consultant, Study Director — jordan university
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
on reasonable request